CLINICAL TRIAL: NCT02583178
Title: A Single-arm, Open Label, Multi-Centre Feasibility Study of the Aegis Sierra Ligation System in Left Atrial Appendage Closure in Patients With Atrial Fibrillation
Brief Title: Feasibility Study of a Left Atrial Appendage Closure Device in Patients With Atrial Fibrillation
Acronym: LASSO-AF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Aegis Medical Innovations (Industry)
Collaborators: Applied Health Research Centre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGS-CLIN-003
Record Dates: First submitted 2015-10-20; First posted 2015-10-22 (Estimated); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Aegis Sierra Ligation System (Experimental): The Aegis Sierra Ligation System is a series of devices designed for epicardial ligation of the Left Atrial Appendage through a minimally invasive transcatheter approach.
  Interventions: Device: Aegis Sierra Ligation System

INTERVENTIONS:
Device: Aegis Sierra Ligation System — The SLS is a series of devices designed for epicardial ligation of the left atrial appendage through a minimally invasive transcatheter approach.
  Other Names: Sierra Ligation System; SLS

SUMMARY:
The purpose of this study is to assess the safety and function of the Aegis Sierra Ligation System in accessing and closing off the left atrial appendage (LAA) using a minimally invasive epicardial access approach.

A minimum of 30 participants will be included in this study, which is being performed at a maximum of 8 centers in Canada and the United States. (A maximum of 15 participants at 4 US centers will be enrolled)

Participants will be considered for this treatment if their doctor(s) have determined they have documented non-valvular atrial fibrillation and are at increased risk for developing a stroke.

DETAILED DESCRIPTION:
Study Purpose:

The objective of this early feasibility study is to assess the safety and function of the Aegis Sierra Ligation System (SLS) in ligating the left atrial appendage in patients with non-valvular atrial fibrillation and at risk for stroke. The results of this trial will be used to inform a larger pivotal trial that will allow for further health technology assessment and for Medical Device License applications.

General Design:

This is a prospective, single-arm, open-label, multi-center study. This study will screen patients with atrial fibrillation at risk for stroke. A minimum of 30 patients that meet all of the study's inclusion criteria, none of the exclusion criteria and consent to study participation will be enrolled. Patient accruement will take place at up to 8 North American centers (A maximum of 15 participants at 4 US centers will be enrolled).

Each subject will undergo the following study visits: Screening, LAA ligation Procedure (Day 0) and Post-procedure, Hospital Discharge, Day 7, Day 30, Day 90, Day 180 and Day 365.

The total duration of participation for subjects is anticipated to be 5 years post ligation procedure with the primary safety outcome assessed at the 30-day follow-up and the secondary endpoints assessed at Days 30, 180 and 365. Subjects will be also be contacted for an annual telephone follow-up evaluation from years 2 through 5 to assess for patient-reported long-term Major Adverse Events (MAE) and current health status.

ELIGIBILITY:
Inclusion Criteria:

1. Age >=18 years
2. Documented non-valvular atrial fibrillation
3. Current CHA2DS2-VASc score of ≥2
4. Have an appropriate rationale to seek a non-pharmacologic alternative to oral anticoagulation (OAC) therapy
5. Willing and able to provide written informed consent
6. Willing and able to comply with study procedures and follow-up visits.
7. Able to take antiplatelet therapy post ligation procedure

Exclusion Criteria:

1. Cardiogenic shock or hemodynamic instability
2. Myocardial infarction in the past 3 months
3. Cerebral embolism, stroke, or TIA in past 3 months
4. Absence of a defined left atrial appendage on echocardiogram or CT scan
5. Previous cardiac surgery involving opening of the pericardium
6. History of pericarditis or pericardial tumor, a history of constrictive pericarditis or features which in the opinion of the investigator are suggestive of constrictive pericarditis
7. History of significant chest trauma of the anterior chest
8. Estimated life expectancy < 24 months
9. Chemotherapy in the past 12 months
10. Prior thoracic radiation therapy
11. Chronic liver disease (greater than Child-Pugh Class A), chronic renal disease/insufficiency/failure (creatinine >3.0 mg/dL and/or renal replacement therapy at the time of screening), or chronic end stage pulmonary disease (FEV1 less than 30% predicted).
12. Current use of long-term treatment with steroids. Does not include intermittent use of inhaled steroids for respiratory diseases.
13. Contraindication to transesophageal echocardiography (TEE).
14. Absolute contraindication to anticoagulation or antiplatelet therapy
15. Congenital Heart Disease or intracardiac/intrapulmonary shunts
16. Symptomatic or known significant carotid disease and/ or aortic arch atheroma
17. Known thrombus in the LAA/LA or thrombus visualized by TEE within 48 hours before procedure
18. Left ventricular ejection fraction (LVEF) below 30%
19. Pregnant, breastfeeding or planning pregnancy within next 12 months
20. Inappropriate appendage morphology (aberrant anatomy) as determined by imaging and assessed by Central Screening Committee
21. Current NYHA Class IV heart failure symptoms
22. Right ventricular dysfunction and /or pulmonary hypertension (>=50mmHG)
23. Moderate or greater valve disease (i.e., MVA <1.5cm2, AVA <1.5cm2), history of rheumatic mitral stenosis, or mechanical valve prosthesis.
24. Cardiac tumour
25. Known hypersensitivity to nickel
26. Patients in whom pericardial access will put the patient at risk (e.g. scoliosis, pectus excavatum, massive obesity with a BMI >40) as determined by clinical site Principal Investigator or Central Screening Committee.
27. Current enrollment in an investigation or study of a cardiovascular device or investigational drug that would interfere with this study.
28. Mental impairment or other conditions, which may not allow patient to understand the nature, significance and scope of the study.
29. Any other criteria, which would make the patient unsuitable to participate in this study as determined by clinical site Principal Investigator or Central Screening Committee (e.g., uncontrolled drug and/or alcohol addiction, extreme frailty).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-08-25 (Actual); Primary Completion 2020-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Number of participants free from the safety composite of device or procedure-related Major Adverse Events | Day 30 from procedure
  Major Adverse Events : (defined as)
  * All-cause death
  * Stroke
  * Systemic embolism
  * Major or life-threatening bleeding (VARC-II definition),
  * Injury to coronary arteries requiring intervention,
  * Myocardial infarction (VARC-II definition),
  * Unplanned operation or interventional procedure for device or procedure related complications (including drainage of pericardial effusion),
  * Complications related to epicardial access

SECONDARY OUTCOMES:
Number of participants that experience a safety composite event | Day 30, 6-months and 1-year from procedure
  Components of the safety composites: All-cause death, stroke, trans-ischemic attack (TIA), systemic embolism
Number of participants that experience all-cause death | Day 30, 6-months and 1-year from procedure
  Number of participants that experience all-cause death at each designated time-point
Number of participants that experience stroke | Day 30, 6-months and 1-year from procedure
  Number of participants that experience stroke at each designated time-point
Number of participants that experience a trans-ischemic attack (TIA) | Day 30, 6-months and 1-year from procedure
  Number of participants that experience TIA at each designated time-point
Number of participants that experience systemic embolism | Day 30, 6-months and 1-year from procedure
  Number of participants that experience systemic embolism at each designated time-point
Number of participants that experience severe pericarditis | Day 30, 6-months and 1-year from procedure
  Number of participants that experience severe pericarditis at each designated time-point
Number of participants that experience worsening heart failure | Day 30, 6-months and 1-year from procedure
  Worsening heart failure is defined as an increase in New York Heart Association (NYHA) Class ≥ category
Number of participants that experience a new occurrence of left atrial thrombus | Day 30, 6-months and 1-year from procedure
  Number of participants that experience a new occurrence of LAA thrombus at each designated time-point
Number of participants that experience an access site wound infection requiring IV antibiotics | Day 30, 6-months and 1-year from procedure
  Number of participants that experience an access site wound infection requiring antibiotics at each designated time-point
Number of participants that achieve Technical Success | Assessed at end of procedure
  Technical success is defined as proper placement and positioning of the device includes the ability to access the pericardium, locate and grasp the LAA, and secure the ligating loop
Number of participants that achieve Procedural Success | Hospitalization period
  Defined as Technical Success and no Major Adverse Events
Number of participants that achieve a residual flow ≤ 5mm distal to the closure site as measured by transesophageal echo (TEE) | Day 30, 6-months and 1-year from procedure
  Number of participants that achieve a residual flow ≤ 5mm distal to the closure site as measured by transesophageal echo (TEE) at each time-point
The reported average change in B-type Natriuretic Peptide (BNP) | Change between baseline and 6-months from procedure
  Reported in picomole/liter (pmol/L)
The reported average change in the rating of atrial fibrillation burden as measured the University of Toronto Atrial Fibrillation Severity Scale (AFSS v. Sept 25, 2014) | Change between baseline to 6-months and 1-year from procedure
  Change in AFSS score between baseline to 6-months and 1-year from procedure will be reported
The reported average change in Health Related Quality of Life scoring as measured by the Atrial Fibrillation Effect on Quality-of-Life Questionnaire (AFEQT v.1.0) | Change between baseline to Day 30, 6-months, and 1-year from procedure
  Change in AFEQT score between baseline, Day 30, 6-months and 1-year from procedure will be reported
The average change in patient reported pain as measured by the Numeric Rating Scale (NRS-11) pain scale. | Change from baseline to hospital discharge, Day 7, and Day 30 from procedure
  Change in NRS pain score between baseline, hospital discharge,Day 7, and Day 30 from procedure will be reported

CONTACTS AND LOCATIONS:
Overall Officials: Sheldon Singh, MD, Principal Investigator — Sunnybrook Health Sciences Centre, Ontario Canada
Locations (7):
- United States (4):
  - Pacific Heart Institute, Santa Monica, California
  - Mayo Clinic, Rochester, Minnesota
  - Mount Sinai Hospital, New York, New York
  - Houston Methodist Research Institute, Houston, Texas
- Canada (3):
  - St. Paul's Hospital - Heart Rhythm Research, Vancouver, British Columbia
  - Victoria Cardiac Arrhythmia Trials, Victoria, British Columbia
  - Sunnybrook Health Sciences Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Undecided